CLINICAL TRIAL: NCT01240187
Title: A Randomized, Open-label, Crossover Study to Demonstrate Bioequivalence Between 6 x2 mg Tablets of Perampanel and a Single 12 mg Tablet of Perampanel in Healthy Subjects
Brief Title: A Study to Demonstrate Bioequivalence Between 6 x 2 mg Tablets of Perampanel and a Single 12 mg Tablet of Perampanel in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2007-E044-037
Record Dates: First submitted 2010-09-23; First posted 2010-11-15 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-05

CONDITIONS: Partial Onset Epilepsy
Keywords: epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel

ARMS (2):
- Experimental 1 (Experimental)
  Interventions: Drug: perampanel
- Experimental 2 (Experimental)
  Interventions: Drug: perampanel

INTERVENTIONS:
Drug: perampanel — Single dose of 6 tablets 2 mg orally
  Arms: Experimental 1
Drug: perampanel — Single dose of 1 tablet 12 mg orally
  Arms: Experimental 2

SUMMARY:
The purpose of this study is to investigate the bioequivalence between 6 x 2 mg tablets and one 12 mg tablet of perampanel in healthy subjects.

DETAILED DESCRIPTION:
A Single Centre, open label, 2-period, 2-sequence crossover bioequivalence study in one group of 28 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects aged between 18-55 years.
* BMI of 18-32 kg/m ^2.
* Willing and able to provide written informed consent.

Exclusion criteria:

* Subjects taking prescribed or over the counter (OTC) medications in 2 weeks prior to screening.
* Subjects on special diets or dietary aids known to modulate drug metabolizing enzymes.
* Subjects who have taken inhibitor of CYP450 within 2 weeks of first dose.
* Subjects who have received any experimental drug in the 12 weeks prior to study drug treatment.
* Subjects with a history of alcohol abuse or who drink more than the recommended number of alcohol units per week.
* Subjects who consume more than five caffeinated beverages per day.
* Subjects who smoke more than 5 cigarettes per day.
* Subjects with a history of drug abuse or who have a positive urine drug screening test.
* Women who do not agree to use two methods of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the pharmacokinetic (PK) profile, safety, and tolerability of 6 x 2-mg tablets of perampanel with a single 12-mg tablet. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr Joanne Collier, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Edinburgh, United Kingdom